CLINICAL TRIAL: NCT02122562
Title: Functional Neuroimaging of the Enhanced Antidepressant Efficacy of Ketamine in a Biologically-Enriched Subgroup
Brief Title: Ketamine Alcohol (in Treatment-Resistant Depression)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mark Niciu (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Mark Niciu, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201906726; 14-M-0085 (Other: National Institutes of Health); 4R00AA024142-02 (NIH)
Record Dates: First submitted 2014-04-23; First posted 2014-04-24 (Estimated); Last update posted 2025-02-26 (Actual); Status verified 2024-08

CONDITIONS: Magnetic Resonance Imaging; Major Depression; Alcoholism
Keywords: Ketamine; Major Depression; NMDA Antagonist
MeSH Terms: conditions — Depressive Disorder, Major; Alcoholism | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Ketamine — Treatment

SUMMARY:
A single subanesthetic dose infusion of the N-methyl-D-aspartate (NMDA) receptor antagonist ketamine has rapid and robust antidepressant effects in patients with treatment-refractory major depressive disorder (TRD). A family history of an alcohol use disorder (Family History Positive, FHP) is one of the strongest identified predictors of an improved antidepressant response to ketamine. Like ketamine, alcohol is a functional NMDA receptor antagonist. FHP is associated with differential response to ketamine, e.g. blunted psychotomimetic side effects. One of the primary mechanistic hypotheses for ketamine's antidepressant action is the acute intrasynaptic release of glutamate from major output neurons, e.g. cortical pyramidal cells. Preliminary clinical studies have demonstrated this acute glutamate "surge" in response to subanesthetic dose ketamine. Based on these findings, the investigators hypothesize that ketamine's enhanced antidepressant efficacy in FHP TRD subjects is, at least in part, attributable to increased glutamate release relative to TRD subjects without a family history of alcohol use disorder (Family History Negative, FHN). To test this hypothesis, the investigators have designed a now two-site, open-label study of 18-55-year-old medically and neurologically healthy, currently moderately-to-severely depressed TRD patients. In total, the investigators plan to recruit 25 FHP and 25 FHN TRD subjects. All subjects must not have a current substance use disorder (except nicotine or caffeine). The experimental portion consists of two phases. The preliminary first phase is a medication taper (if needed) and psychotropic medication-free period. The experimental second phase comprises one subanesthetic dose (0.5mg/kg x 40 minute) ketamine infusion. The ketamine infusion will occur during 7T-magnetic resonance imaging (MRI), both resting-state functional MRI (rs-fMRI) and magnetic resonance spectroscopy (MRS) to detect glutamate in the ventromedial prefrontal cortex/ventral anterior cingulate cortex (vmPFC/vACC). The primary outcome measure is group mean change in Montgomery-Åsberg Depression Rating Scale (MADRS) score from pre-ketamine infusion (baseline) to one-week post-infusion, where the investigators observed ketamine's greatest antidepressant effect in FHP TRD. Additional outcome measures are vmPFC/vACC glutamate change in response to ketamine based on family history status. In summary, this study will provide key mechanistic information on ketamine's improved antidepressant efficacy in a biologically-enriched subgroup. This will contribute to the systematic development of more efficacious, personalized treatments for major depression in an effort to reduce its enormous public health burden.

DETAILED DESCRIPTION:
Objective:

Glutamate-based medications including the glutamate modulator ketamine result in rapid, robust and sustained (typically up to one week) antidepressant effects in randomized controlled trials in treatment-refractory unipolar and bipolar depression. Previous work by the investigators' group has demonstrated that a family history of alcohol dependence predicts a more robust antidepressant response to ketamine in both treatment-resistant unipolar and bipolar depression.

Recently-detoxified alcoholics and affected first-degree relatives display blunted psychotomimetic, cognitive and other neuropsychiatric effects when administered a subanesthetic dose of ketamine. Based on the prior post hoc results, the investigators seek to prospectively demonstrate that a family history of an alcohol use disorder predicts a more robust antidepressant response to ketamine.

Study Population:

18-55 year old TRD without psychotic features patients in a current major depressive episode of at least moderate severity will be recruited and enrolled in this study. All subjects must not have a current substance use disorder (except nicotine or caffeine). All subjects must be psychotropic medication-free for at least two weeks prior to the ketamine infusion. The targeted number of completers is 50 depressed subjects (60 signing consent to account for attrition): 25 FHP subjects [as defined by either one first degree relative or two second-degree relatives with an alcohol user disorder on the Family Interview for Genetics Studies (FIGS) and Family Tree Questionnaire (FTQ)] and 25 FHN negative subjects.

Design:

This study is currently a single site, open-label protocol in psychotropic medication-free depressed subjects. This protocol consists of two phases. Phase I consists of a medication taper (if needed) and at least two week drug-free period. Phase II includes a subanesthetic/antidepressant dose ketamine infusion during 7T-MRI.

Outcome Measures:

The primary hypothesis/outcome measure will be mean change in MADRS total score from the pre-ketamine infusion (baseline) to 7 days post-infusion between the FHP and FHN groups. Other exploratory measures include glutamate alterations during intravenous ketamine infusions and rs-fMRI as a function of family history status.

ELIGIBILITY:
INCLUSION CRITERIA:

1. 18 to 55 years of age.
2. A level of understanding sufficient to agree to all required tests and examinations, sign an informed consent document and verify understanding by a score greater than or equal to 90% on the consent quiz.
3. Diagnostic and Statistical Manual-4th Edition-Text Revision (DSM-IV-TR)) diagnosis of major depressive disorder (MDD), single-episode (296.30) or recurrent (296.20) without psychotic features based on clinical assessment and confirmed by a Structured Clinical Interview for the DSM-IV- Patient Version (SCID-P). Subjects must be experiencing a current major depressive episode of at least 2 weeks duration.
4. Past failure of greater than or equal to one standard antidepressant trial based on the Antidepressant Treatment History Form (ATHF).
5. MADRS score greater than or equal to 20 at baseline and the day of ketamine infusion.

EXCLUSION CRITERIA:

1. Inadequate knowledge of family mental and substance use history, e.g. adoption.
2. Current psychotic features or prior diagnosis of a DSM-IV-TR psychotic spectrum disorder, e.g. schizophrenia, schizoaffective disorder, bipolar I disorder with psychotic features, MDD with psychotic features, or bipolar disorder, e.g. bipolar I disorder without psychotic features, bipolar II disorder and bipolar disorder not otherwise specified (NOS).
3. Current/active DSM-IV-TR substance use disorder (except for caffeine or nicotine dependence).
4. Pregnant or nursing women or women of childbearing potential not using at least one medically accepted means of contraception (to include oral, injectable, or implant birth control, condom or diaphragm with spermicide, intrauterine devices (IUD), tubal ligation, abstinence or partner with vasectomy).
5. Serious, unstable medical conditions/problems including hepatic, renal, gastroenterologic, respiratory, cardiovascular, endocrinologic, neurologic, immunologic, or hematologic disease, e.g. uncontrolled asthma, uncontrolled hyper/hypothyroidism or active cancer.
6. Presence of any medical illness likely to alter brain morphology and/or physiology (e.g., hypertension, diabetes) even if controlled by medications.
7. Clinically significant abnormal laboratory tests.
8. Subjects with one or more seizures without clear and resolved etiology and head injury with loss of consciousness for > 5 minutes or requiring hospitalization.
9. Treatment with psychiatric medications, e.g. selective serotonin reuptake inhibitors, serotonin norepinephrine reuptake inhibitors, benzodiazepines and antipsychotics, at least two weeks of study phase II.
10. Treatment with fluoxetine within 5 weeks of study phase II.
11. Treatment with device-based treatment for depression, e.g. electroconvulsive therapy (ECT), transcranial magnetic stimulation (TMS) and vagal nerve stimulation (VNS), within 4 weeks of study phase II.
12. Lifetime history of deep brain stimulation.
13. Treatment with any disallowed concomitant medications.
14. Positive HIV test
15. Presence of ferromagnetic implants, e.g, heart pacemaker or aneurysm clip, or other contraindications to magnetic resonance imaging (MRI), e.g. claustrophobia or hearing loss.
16. Clinically-significant anatomical brain abnormalities detected on routine brain MRI.
17. Subjects who, in the investigator's judgment, pose a current serious suicidal or homicidal risk, or who have a MADRS item 10 score of greater than or equal to 4.
18. A current NIMH employee/staff or their immediate family member (N.B. former exclusion criteria likely to be no longer relevant at the University of Iowa Health Care).
19. Currently engaged in an evidence-based structured psychotherapy for mood and/or anxiety disorders, e.g. cognitive-behavioral therapy (CBT) or interpersonal psychotherapy (IPT).

Additionally, the investigators may exclude or terminate any patient for clinical reasons.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-04-23; Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) | Pre-ketamine (baseline) to one week post-ketamine infusion
  The MADRS contains 10 items, and each item is scored 0-6. These item scores are summed to create a scale score; thus, scale scores range from 0 to 60. A scale score of 0 indicates the absence of depressive symptoms, while a score of 60 indicates severe depression. The primary outcome is the mean change in total MADRS score. A decrease in the mean MADRS score indicates a decrease (or improvement) in depressive symptoms, whereas an increase in the mean MADRS score indicates an increase (or worsening) in depressive symptoms.

SECONDARY OUTCOMES:
Concentration of Glutamate and Other Neurometabolites | Prior to and during ketamine infusions
  High-magnetic field strength (7T) proton magnetic resonance spectroscopy (1H-MRS) detectable glutamate and other neurometabolites, e.g. N-acetylaspartate and creatine
Resting State Functional Connectivity | Prior to and during ketamine infusions
  Task-free ("resting state") functional magnetic resonance imaging (rs-FMRI) to detect changes in blood oxygen-level dependent (BOLD) signal
Hamilton Depression Rating Scale (HDRS) | Pre-ketamine (baseline) to one week post-ketamine infusion
  The HDRS is a clinician-administered depression rating scale that contains 21 items. The first 17 items are summed to create a total scale score. Score ranges indicate depression severity: 0-7 indicates the absence of depression, 8-13 indicates mild depression, 14-18 indicates moderate depression, 19-22 indicates severe depression, and >22 indicates very severe depression.
Beck Depression Inventory (BDI) | Pre-ketamine (baseline) to one week post-ketamine infusion
  The BDI is a self-administered 21-item measure of depression severity. Each item is scored (in increasing severity) on a scale from 0-3. Total scores range from 0-63: 0-9 indicates no depression, 10-18 indicates mild depression, 19-29 indicates moderate depression, >29 indicates severe depression.
Hamilton Psychiatric Rating Scale for Anxiety (HAM-A) | Pre-ketamine (baseline) to one week post-ketamine infusion
  The HAM-A is a clinician-administered scale of anxiety severity that comprises 14 items rated on a scale of 0-4. The HAM-A total score is the sum of 14 items with a score range from 0-56, with lower scores indicating low levels of anxiety and higher scores indicating greater anxiety severity.
Young Mania Rating Scale (YMRS) | Pre-ketamine (baseline) to one week post-ketamine infusion
  The YMRS scale is an 11-item clinician-administered rating scale to assess hypo/manic symptoms. Items 5, 6, 8, and 9 (irritability, speech, content and disruptive-aggressive behavior) are rated on a scale from 0 (symptom not present) to 8 (symptom extremely severe). The remaining items are rated on a scale from 0 (symptom not present) to 4 (symptom extremely severe). Items 5, 6, 8, and 9 are given twice the weight of the remaining 7 items. The YMRS total score ranges from 0 to 60. Lower scores indicate absence of manic-like symptoms while higher scores indicate increasingly severe manic-like symptoms.
Snaith-Hamilton Pleasure Scale (SHAPS) | Pre-ketamine (baseline) to one week post-ketamine infusion
  The SHAPS scale is a 14-item self-reported instrument to measure anhedonia. Scale scores are created by summing each item. Higher scale scores indicate more anhedonia, and lower scale scores indicate increased hedonic value.
Temporal Experience of Pleasure Scale (TEPS) | Pre-ketamine (baseline) to one week post-ketamine infusion
  The TEPS scale is an 18-item self-reported questionnaire that measures pleasure associated with the consumption and anticipation of rewards. Lower scores indicate less pleasure while higher scores indicate greater hedonic value.
Scale for Suicidal Ideation (SSI) | Pre-ketamine (baseline) to one week post-ketamine infusion
  The SSI is a 19-item clinician-administered instrument designed to quantify the intensity of current conscious suicidal ideation in various dimensions of self-destructive thoughts or wishes: the extent of the wish to die, the desire to make an actual suicide attempt, and details of any plans; also, internal deterrents to an active attempt, and subjective feelings of control and/or courage regarding a proposed attempt. We will administer both the full and a short (5-item) version to assess rapid change in suicidal thinking. Scale scores are calculated by summing item scores and range from 0-38. Lower scores indicate less suicidal ideation and higher scores indicate escalating severity of suicidal thinking.
Columbia-Suicide Severity Rating Scale (C-SSRS) | Pre-ketamine (baseline) to one week post-ketamine infusion
  The C-SSRS is a clinician-administered instrument designed to measures suicidal ideation/behaviors with both "Lifetime/Recent" and "Since Last Visit" versions. There are four subscales. Severity of ideation subscale is measured on a 5-point ordinal scale in which 1=wish to be dead, 2=nonspecific active suicidal thoughts, 3=suicidal thoughts with methods, 4=suicidal intent, and 5=suicidal intent with plan. The intensity of ideation subscale has 5 items: frequency, duration, controllability, deterrents, and reason for ideation, which is rated on a 5 point scale. The suicidal behavior subscale is rated on attempts, preparatory behavior, and nonsuicidal self-injury. The lethality subscale measures lethalities of actual attempts, which is rated on a 6 point scale.
Alcohol Urge Questionnaire (AUQ) | Pre-ketamine (baseline) to one week post-ketamine infusion
  The AUQ is an 8-item self-report scale to assess acute alcohol cravings. It utilizes a 7 point Likert scale, and items are summed for a total scale score, where higher scores indicate greater cravings/urges to drink alcohol. This measure will be used to assess alcohol-related expectancies with both alcohol and ketamine.
Obsessive Compulsive Drinking Scale (OCDS) | Pre-ketamine (baseline) to one week post-ketamine infusion
  The OCDS is a self-administered instrument that consists of 14 items that has been shown to be sensitive and specific for the obsessive and compulsive characteristics of alcohol misuse: drinking-related preoccupations, urges to drink, and the ability to desist these thoughts/urges. This measure will also be used to assess alcohol-related expectancies related to both alcohol and ketamine infusions. Items are rated on a 5 point Likert scale. Higher scores indicate more preoccupation, urges, or difficulty controlling urges to drink/consume alcohol.
Brief Psychiatric Rating Scale (BPRS) | Pre-ketamine (baseline) to one week post-ketamine infusion
  The BPRS is a clinician-administered instrument with 4 key items will be used as an index of positive symptoms of schizophrenia. These 4 key positive domains are conceptual disorganization, hallucinatory behavior, suspiciousness and unusual thought content. 3 additional BPRS items - blunted affect, emotional withdrawal and motor retardation - are selected as a measure of negative schizophrenia symptoms. Each item is scored on a 7 point Likert scale, with 1 indicating absence of a given symptom and 7 indicating highest measured severity. Individual item are added to form a total scale score.
Visual Analog Scale (VAS) | Pre-ketamine (baseline) to one week post-ketamine infusion
  The VAS is a 7-item self-administered Likert-type measure with individual items scored between 0-10. This instrument rates 7 domains: happy/euphoric, restless, sad, anxious, irritated/angry, drowsy and alert. A score of 0 is described as "none", 1-3 is "mild", 4-6 is "moderate", 7-9 is "marked" and 10 is "extreme" for each given item.
Clinician-Administered Dissociative States Scale (CADSS) | Pre-ketamine (baseline) to one week post-ketamine infusion
  The CADSS is a measure of perceptual, behavioral and attentional changes occurring during dissociative experiences that has been tested in healthy subjects and post-traumatic stress disorder (PTSD). This scale involves 19 self-reported questions and 8 observer ratings scored from 0 (not at all) - 4 (extremely). Greater scores indicate greater ketamine-induced dissociation.
Clinical Global Impression/Severity (CGI) | Pre-ketamine (baseline) to one week post-ketamine infusion
  The CGI is a clinician-measured scale of 3 items: Severity of Illness (item 1), Global Improvement (item 2), and Efficacy Index (item 3). Items 1 and 2 are rated on a 7-point Likert scale (1=normal, 7=among the most extremely ill patients) with a possible response of "not assessed." Item 3 is rated on a 4-point Likert scale from "none" to "outweighs therapeutic effect." Items 1 and 3 are assessed in relation to last clinical encounter (if possible).
Modified Version of the NIMH Data Safety Event Codes (NIMH-DSEC) | Pre-ketamine (baseline) to one week post-ketamine infusion
  This clinician-collected form collects information over 100 symptoms/signs across multiple organ systems. The "Specific" form is for tracking side effects that are often seen during the infusion at multiple time points. The "Regular" form is for the baseline (-60 minutes), +230 minute post-ketamine infusion (final time point on the day of ketamine infusion) and other daily time points post-ketamine infusion.
The Positive and Negative Affect Schedule (PANAS) | Pre-ketamine (baseline) to one week post-ketamine infusion
  The PANAS is a self-report questionnaire comprised of 2 mood scales, one that measures positive affect and one that measures negative affect. Used as a psychometric scale, the PANAS can show relations between positive and negative affect with personality states and traits. 10 descriptors are used for each positive and negative affect scale to define their meanings. Participants are asked to respond to a 20-item test, and each individual item is scored on a a 5-point Likert scale that ranges from very slightly or not at all (1) to extremely (5).

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Niciu, M.D. Ph.D., Principal Investigator — University of Iowa Health Care (UIHC)
Locations (1):
- University of Iowa Health Care, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berman RM, Cappiello A, Anand A, Oren DA, Heninger GR, Charney DS, Krystal JH. Antidepressant effects of ketamine in depressed patients. Biol Psychiatry. 2000 Feb 15;47(4):351-4. doi: 10.1016/s0006-3223(99)00230-9. PMID 10686270
- [Background] Zarate CA Jr, Singh JB, Carlson PJ, Brutsche NE, Ameli R, Luckenbaugh DA, Charney DS, Manji HK. A randomized trial of an N-methyl-D-aspartate antagonist in treatment-resistant major depression. Arch Gen Psychiatry. 2006 Aug;63(8):856-64. doi: 10.1001/archpsyc.63.8.856. PMID 16894061
- [Background] Valentine GW, Mason GF, Gomez R, Fasula M, Watzl J, Pittman B, Krystal JH, Sanacora G. The antidepressant effect of ketamine is not associated with changes in occipital amino acid neurotransmitter content as measured by [(1)H]-MRS. Psychiatry Res. 2011 Feb 28;191(2):122-7. doi: 10.1016/j.pscychresns.2010.10.009. Epub 2011 Jan 12. PMID 21232924